CLINICAL TRIAL: NCT03631914
Title: Intelligent Needle Tip Tracking Using Ultrasound Imaging for Infraclavicular Brachial Plexus Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Philips Medical Systems (Industry); B. Braun Melsungen AG (Industry)
Responsible Party: Principal Investigator, Axel Rudolf Sauter, Pricipal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2018/1098
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Nerve Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active needle tip tracking (Active Comparator): A needle tip tracking system is used when performing an ultrasound guided infraclavicular brachial plexus block.
  Interventions: Procedure: Infraclavicular brachial plexus block
- Inactive needle tip tracking (Other): No needle tip tracking system is used when performing an ultrasound guided infraclavicular brachial plexus block.
  Interventions: Procedure: Infraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Infraclavicular brachial plexus block — An infraclavicular brachial plexus block is performed using ultrasound guidance.

SUMMARY:
In a randomized controlled crossover study design, ultrasound guided infraclavicular brachial plexus blocks will be performed with and without the aid of a needle tip tracking (NTT) system. Specialists in anaesthesiology with average experience in ultrasound guided PNB techniques will perform the blocks. 26 volunteers will be included. The primary objective is to investigate the effect of the NTT system on performance time, as a measure for improved block performance. Secondary objectives are the effects of the NTT system on dexterity, peripheral nerve block characteristics, subjective experience, and peripheral block performance.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2
* Volunteers that have given informed written consent

Exclusion Criteria:

* BMI < 18 kg/m2
* BMI > 35 kg/m2
* Body weight > 95 kg
* Volunteers that cannot cooperate during the examination
* Volunteers that do not speak or understand Norwegian language
* Volunteers with neurologic disease, nerve- or vascular impairment
* Volunteers with known coagulopathy
* Volunteers that are allergic to Lidocaine or other local anaesthetic agents
* Medications at the investigators discretion
* Volunteers with concomitant medical treatments interfering with PNB treatment
* Skin disease or infection affecting the whole-body surface or within the area of examination
* Any reason why, in the opinion of the investigators, the volunteer should not participate
* Subject participates in a potentially confounding drug or device trial during the course of the study
* Pregnancy and lactation period
* Women of childbearing potential who do not use an effective and secure method for birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Performance time | During peripheral nerve block procedure
  Performance time is defined as the time from insertion of the block needle (skin puncture) until finishing LA injection

SECONDARY OUTCOMES:
Distance travelled by needling hand | During peripheral nerve block procedure
  Measured by motion analysis from insertion of the block needle (skin puncture) until finishing LA injection
Distance travelled by probe hand | During peripheral nerve block procedure
  Measured by motion analysis from insertion of the block needle (skin puncture) until finishing LA injection
Number of intended movements (needling hand) | During peripheral nerve block procedure
  Measured by motion analysis from insertion of the block needle (skin puncture) until finishing LA injection
Number of intended movements (probe hand) | During peripheral nerve block procedure
  Measured by motion analysis from insertion of the block needle (skin puncture) until finishing LA injection
Block success | 30 minutes after peripheral nerve block procedure
  A sensory block is defined as successful when there is analgesia (no sensation for touch) or anaesthesia (no sensation at all) involving all five nerves distal to the elbow
Block onset time | Within 60 minutes after peripheral nerve block procedure
  Block onset time is defined as the time between the end of LA injection and development of a successful sensory block
Block duration | Within 240 minutes after peripheral nerve block procedure
  Block duration is the time from the end of LA injection until at least one of the nerves involved in the sensory block has recovered
Quantified discomfort during block performance | Immediately after peripheral nerve block procedure
  The participants are asked about discomfort during the block procedure using a numeric rating scale (scale range 0 - 10; 0 = no discomfort; 10 = worst discomfort imaginable)
Confidence in block success | Immediately after peripheral nerve block procedure
  The anaesthetist is asked if he expects the block to be successful using a numeric rating scale (scale range 0 - 10; 0 = block success unlikely; 10 = block success very likely)

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Kasine T, Romundstad L, Rosseland LA, Fagerland MW, Kessler P, Omenas IN, Holmberg A, Sauter AR. Ultrasonographic needle tip tracking for in-plane infraclavicular brachialis plexus blocks: a randomized controlled volunteer study. Reg Anesth Pain Med. 2020 Aug;45(8):634-639. doi: 10.1136/rapm-2020-101349. Epub 2020 Jun 14. PMID 32540878